CLINICAL TRIAL: NCT02656147
Title: Phase I Study of γδT Cells Expressing an Anti-CD19 Chimeric Receptor in Children and Young Adults With B Cell Malignancies
Brief Title: Immunotherapy With CD19 CAR γδT-cells for B-Cell Lymphoma, ALL and CLL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Doing Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doing-004
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; CAR γδT
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: 1 (Experimental): Acute lymphoblastic leukemia treated with chimeric antigen receptor modified γδT cells(Anti-CD19-CAR γδT) targeting CD19.
  Interventions: Biological: Anti-CD19-CAR γδT
- Experimental: 2 (Experimental): Chronic lymphoblastic leukemia with chimeric antigen receptor modified γδT cells(Anti-CD19-CAR γδT) targeting CD19.
  Interventions: Biological: Anti-CD19-CAR γδT
- Experimental: 3 (Experimental): Non-hodgkin lymphoma treated with chimeric antigen receptor modified γδT cells(Anti-CD19-CAR γδT) targeting CD19.
  Interventions: Biological: Anti-CD19-CAR γδT

INTERVENTIONS:
Biological: Anti-CD19-CAR γδT — Cells extracted, followed by induction chemotherapy before Anti-CD19-CAR γδT infusion (dose escalation.)

SUMMARY:
This study aims to evaluate the safety, efficacy and duration of response of CD19 Chimeric Antigen Receptor (CAR) redirected allogeneic γδT-cells in patients with high risk, relapsed CD19+ haematological malignancies.

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product named CD19 Chimeric Antigen Receptor (CAR) γδT-cells (CD19 CAR γδT-cells) in patients with high risk, relapsed CD19+ haematological malignancies (Leukemia and lymphoma). Following informed consent and registration to the trial, Patients will receive the allogeneic CD19 CAR γδT-cells following lymphodepleting chemotherapy. The study will evaluate the safety, efficacy and duration of response of the CD19 CAR γδT-cells in patients with high risk relapsed CD19+ malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory B cell derived acute lymphoblastic leukemia(ALL), chronic lymphoblastic leukemia(CLL) and non-hodgkin lymphoma.
2. KPS>60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 18 years to 70 years.
5. CD19 expression must be detected on greater than 15% of the malignant cells by immunohistochemistry or greater than 30% by flow cytometry.
6. Patients who have failed at least one line of a standard treatment.
7. No serious mental disorder.
8. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
9. No other serious diseases(autoimmune disease, immunodeficiency etc.).
10. No other tumors.
11. Patients volunteer to participate in the research.
12. Patients with history of allogeneic stem cell transplantation are eligible if at least 100 days post-transplant, if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to infusion.

Exclusion Criteria:

1. KPS<50.
2. Patients are allergic to cytokines.
3. Central nervous system leukemia within 28 days.
4. Uncontrolled active infection.
5. Acute or chronic GVHD.
6. Treated with T cell inhibitor.
7. Pregnancy and nursing females.
8. HIV/HBV/HCV Infection.
9. Other situations we think improper for the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events of each patient. | 3 years
  Adverse events of each patient will be recorded and analysed.

SECONDARY OUTCOMES:
Survival time of Anti-CD19 CAR γδT cells in vivo. | 3 years
  PCR will be applied to analyse the survival time of Anti-CD19 CAR γδT cells in vivo.
Antitumor Effects | Every 3 months post treatment up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.
Maximum tolerated dose (MTD) of CD19 targeted CAR γδT cells. | 4 weeks
  Maximum tolerated dose (MTD) of CD19 targeted CAR γδT cells.

CONTACTS AND LOCATIONS:
Overall Officials: Li gangyi, master, Study Chair — Beijing Doing Biomedical Co., Ltd.
Locations (1):
- Beijing DOING Biomedical Co., Ltd, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided